CLINICAL TRIAL: NCT03189407
Title: Evaluation of the Effect of Moringa Oleifera Tea on Metformin Steady State Plasma Level in Type 2 Diabetes Mellitus Patients - a Pre and Post Non-randomised Trial
Brief Title: Effect of Moringa Oleifera on Metformin Plasma Level in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Titilayo O Fakeye (Other)
Responsible Party: Sponsor-Investigator, Titilayo O Fakeye, Professor, University of Ibadan
Organization: University of Ibadan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHI001
Record Dates: First submitted 2017-06-05; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Moringa Oleifera tea; Type 2 Diabetes Mellitus; Metformin Steady state concentrations; Herb-drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moringa oleifera tea in T2DM patients (Other): The study was a pre/post design for type 2 diabetes mellitus patients on metformin in which each patient acted as his/her control. Intervention of twice daily pre-packed 400g dried Moringa oleifera leaves to be prepared as tea by the patients was done. Evaluation of the effect of the tea on metformin steady state concentrations and blood glucose measurements were done.
  Interventions: Dietary Supplement: Moringa oleifera tea

INTERVENTIONS:
Dietary Supplement: Moringa oleifera tea

SUMMARY:
Type 2 diabetes mellitus (T2DM) patients from our previous survey tend to co-administer various herbs with their oral hypoglycemic agents (OHA). Some of these herbs are known to possess antidiabetic activities. One of such is Moringa oleifera leaves.

The present study evaluated the effects of seven days, twice-daily administration of hot water infusion of dried Moringa oleifera leaves on the steady state plasma concentrations of Metformin, one of the most widely used OHAs using T2DM patients who have been on Metformin for a period of not less than three months. The included patients had also been on Moringa supplementation but had terminated the use of Moringa at least a month to the start of the study.

Patients who had other comorbidities such as heart diseases, renal or hepatic impairments were excluded from the study. The patients were recruited from Endocriniology clinic of the Obafemi Awolowo University Teaching Hospitals complex, a tertiary hospital from southwest Nigeria.

Each patient served as his/her control.

DETAILED DESCRIPTION:
Background Plant parts of Moringa oleifera Lam. (Moringaceae) is known to lower blood glucose level and as a result, type 2 diabetes mellitus patients (T2DM) sometimes use it as herbal supplements. This study therefore sought to evaluate the effects of coadministration of Moringa oleifera tea on steady state concentration of metformin in ambulatory T2DM patients attending a tertiary health facility in Nigeria.

Method This study used a non-randomized pre-test and post-test design to evaluate the effects of coadministration of Moringa tea and metformin on selected parameters in T2DM patients. Consented patients, aged 49 -77 years were stabilised on the same brand of metformin for seven days. On day 8 after an overnight fast, baseline fasting blood sugar (FBG) and 2-hour post prandial blood sugar (2-hPPBG) were determined using a glucometer. Blood samples were also collected at the appropriate times for evaluation of serum creatinine, trough and peak metformin plasma concentrations.

Thereafter, patients were given fourteen sachets of pre-packed 400 g dried Moringa oleifera leaves for preparation of Moringa tea for seven days (twice daily) while on their normal doses of metformin. On day 15 after an overnight fast, a repeat of FBG and 2-hPPBG was done using a glucometer. At the appropriate times, blood samples were also collected for determination of serum creatinine, trough and peak metformin plasma concentrations.

Serum was obtained from aliquots of the blood samples to determine serum creatinine for calculation of estimated glomerular filtration rate, eGFR. Plasma was obtained from the blood samples and were analysed using modified previously-validated HPLC method.

The values of FBG, 2-hPPBG, trough and peak metformin plasma concentrations obtained were compared with the baseline values using Paired sample t-test at P<0.05 considered significant in order to evaluate the effect of Moringa tea on the parameters.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory type 2 diabetes mellitus patients from 40 years of age who had supplemented their oral hypoglycaemic drugs with Moringa oleifera in the past but had stopped for over one month were recruited into the study.

Exclusion Criteria:

* Patients with co-morbidities such as congestive heart failure, liver disease, and those who had undergone recent surgical procedure were excluded from the study. Other types of patient excluded from the study were: patients on insulin or whose oral hypoglycaemic drug therapy does not include metformin, patients who take alcohol, patients who were on cimetidine, furosemide, nifedipine, ciprofloxacin, rifampicin, anti-retroviral therapy or any other medication with known interactions with metformin. Patients who smoked were also excluded.

Ages: 49 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Blood Glucose | Change from Baseline Fasting Blood Glucose at 1 week
  Blood glucose (mmol/L) after overnight fast after 7-day Moringa tea, with continuous use of metformin
Change in Two-hour Post Prandial Blood Glucose | Change from Baseline Two-hour Post Prandial Blood Glucose at 1 week
  Blood glucose (mmol/L) two hours after breakfast after 7-day Moringa tea, with continuous use of metformin
Change in metformin trough plasma concentration | Change in metformin trough concentration at 1 week
  Plasma level of metformin (ug/mL) pre-dose in the morning after 7-day Moringa tea, with continuous use of metformin
Change in metformin peak plasma concentration | Change in metformin peak concentration at 1 week
  Plasma level of metformin (ug/mL) two hours post dose after 7-day Moringa tea, with continuous use of metformin
Change in estimated glomerular filtration rate | Change in estimated glomerular filtration rate at 1 week
  Calculation of glomerular filtration rate (mL/min) from serum creatinine level, pre and post 7-day Moringa tea supplementation and continuous use of metformin

CONTACTS AND LOCATIONS:
Overall Officials: Toyin Famurewa, B.Pharm;MSc, Principal Investigator — Obafemi Awolowo University Hospitals Complex, Ile-Ife, Nigeria

IPD SHARING:
Plan to Share IPD: No
The data will only be made public as a publication in a peer-reviewed journal. Also, the Endocrinologist in the team is aware of the results obtained and the implications of using Moringa tea on therapy outcome for a patient on metformin